CLINICAL TRIAL: NCT06774118
Title: Evaluation of Chest Wall Motion Symmetry During Ventilation in Healthy Subjects by Optoelectronic Plethysmography
Acronym: EVAST
Status: Not yet recruiting | Type: Observational
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2024_RIPH_21_EVAST
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Ventilation
Keywords: breathing symmetry; optoelectronic plethysmography; pulmonary ventilation
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy subjects: Consenting healthy subjects with no previous major surgical, traumatic or medical cardiopulmonary history.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
Pulmonary ventilation is the only macroscopically observable breathing step. The ventilatory mechanism has been extensively studied and knowledge of its operation is now well established. The thoraco-abdominal couple is generally considered as a homogeneous functional unit. The anatomical organization of the trunk is not symmetrical. The right lung receives 55% of the volume of air mobilized, the heart is usually lateralized to the left and exerts a mechanical stress on the left lung, the thoracic diaphragm is asymmetrical. The densities of the subdiaphragmatic viscera vary greatly between hollow organs (stomach, colon) and full organs (liver rate).

Conventional spirometry, the gold-standard reference method in ventilatory analysis, allows to measure the quantities of air mobilized at inspiration and expiration. This quantitative method does not provide information on the kinematics of the different areas of the thorax and abdomen involved during breathing.

Optoelectronic plethysmography (OEP) is a non-invasive technique for the analysis of the 3D motion of passive markers placed on the surface of the subject's chest, abdomen and back. This technique, validated as a reliable alternative to conventional spirometry, allows the combination of quantitative measurements of respiratory volumes with qualitative measurements of thoraco-abdominal kinematics. The OEP has the specificity of allowing to choose a segmentation of the trunk to analyze the kinematics of the different identified zones. The most commonly used method in research is segmentation into three compartments (pulmonary thoracic, abdominal and abdominal thoracic).

The OEP studies also suggested the use of segmentation in relation to the median plane of the body to compare the symmetry of the three compartments described above. This 6-compartment segmentation was rarely used in respiratory analysis to assess interventions such as surgery of pulmonary rehabilitation protocols. To our knowledge, there is no study in healthy subjects to assess the level of symmetry of pulmonary ventilation. This type of study is a fundamental preliminary step to be able to subsequently study the symmetry of the ventilatory kinematics in the case of pathologies giving deformities of the thorax, spine and abdomen (scoliosis for example).

DETAILED DESCRIPTION:
The main objective is to describe the degree of symmetry of the ventilatory kinematics in a healthy population using optoelectronic plethysmography to study thoracoabdominal-kinematics in a non-invasive manner by using a 3D optoelectronic motion analysis system in healthy subjects using a 6-compartment digital decomposition.

ELIGIBILITY:
Inclusion Criteria:

* aged between 10 and 70
* with no prior major cardiopulmonary surgical, traumatic or medical history
* agreeing to participate in the study

Exclusion Criteria:

* A major medical cardiopulmonary history, or a history of surgery or trauma to the thorax, abdomen or spine.
* A major medical cardiopulmonary history included any pathology requiring hospital treatment or allopathic therapy lasting more than 3 months.
* Active smoker
* Protected by law (guardianship, curatorship, safeguard of justice)
* Refusing to take part in the study

Ages: 10 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of consenting healthy subjects over 10 years of age, with no major surgical, traumatic or medical cardiopulmonary antecedents.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
pulmonary ribcage asymmetry score | Day 0
  Opto-electronic plethysmography (OEP), using a 3D motion analysis system consisting of 8 optitrack FLEX 13 cameras and 93 passive markers placed on the thorax, abdomen and back of the subject, will assess the volume of all 6 compartments (pulmonary ribcage, abdominal ribcage and their subdivision into left and right parts).
  pulmonary chest asymmetry score will be the difference between the volume of pulmonary ribcage right and the volume of pulmonary ribcage left

SECONDARY OUTCOMES:
abdominal ribcage asymmetry score | Day 0
  Opto-electronic plethysmography (OEP), using a 3D motion analysis system consisting of 8 optitrack FLEX 13 cameras and 93 passive markers placed on the thorax, abdomen and back of the subject, will assess the volume of all 6 compartments (pulmonary ribcage, abdominal ribcage and right and left abdomen).
  abdominal chest asymmetry score will be the difference between the volume of abdominal ribcage right and the volume of abdominal ribcage left
abdominal ribcage asymmetry score | Day 0
  Opto-electronic plethysmography (OEP), using a 3D motion analysis system consisting of 8 optitrack FLEX 13 cameras and 93 passive markers placed on the thorax, abdomen and back of the subject, will assess the volume of all 6 compartments (pulmonary ribcage, abdominal ribcage and right and left abdomen).
  abdomen asymmetry score will be the difference between the volume of abdomen right and the volume of abdomen left

IPD SHARING:
Plan to Share IPD: Undecided